Y Protocol



# Sohag University Faculty of Medicine Department of Rheumatology & Rehabilitation



# Comparison of clinical and serological differences among juvenile, adult, and late-onset systemic lupus erythematosus

#### **Protocol**

Submitted for fulfillment for the requirement of the M.D. Degree in Physical Medicine, Rheumatology and Rehabilitation

# By Alaa Mohamed Hemdan

Assistant lecture of Physical Medicine, Rheumatology and Rehabilitation, Faculty of Medicine, Sohag University

## **Supervised by**

# Dr. Esam Mohamed Abu Al-Fadl

Professor of Physical Medicine, Rheumatology and Rehabilitation Faculty of Medicine, Sohag University

# Dr.Hanan Sayed Mohamed Abo Zaid

Assistant Professor of Physical Medicine, Rheumatology and Rehabilitation Faculty of Medicine, Sohag University

> Faculty of Medicine Sohag University 2022

## **Introduction**

Systemic lupus erythematosus (SLE) is a heterogeneous autoimmune disease with a highly variable presentation and course. It can affect virtually every organ of the body and many symptoms may be observed. Skin, musculoskeletal, hematologic, and serological involvement are most commonly observed. [1] Some patients show predominately hematologic, renal, or central nervous system manifestations. [2,3]

The presentation of SLE may be characterized by periods of remission and by chronic or acute relapses. Several factors, including age and ethnicity, can affect the course and severity of SLE and response to treatment varies by race, ethnicity, and age. Non-Caucasians tend to exhibit acute disease onset, more severe and numerous clinical manifestations, and higher disease activity.[4–10] Hispanics, African descendants and Asians exhibit more frequent renal, hematological, serosal, neuropsychiatric and immunological abnormalities.[5,7,11–14] Furthermore, response to treatment for lupus nephritis varies according to race and ethnicity.[15] Similarly, ethnicity can affect the nature and severity of SLE and its response to treatment: Age of onset also influences the clinical manifestations and severity of SLE. Approximately 15–20% of SLE patients experience disease onset before to adulthood, and about 2–20% of all patients with SLE experience onset of SLE after age of 50.[16–18]

Studies have reported that juvenile-onset SLE patients tend to have a more aggressive presentation and course, with higher rates of organ involvement and lower life expectancy than adult-onset SLE patients.

[19–24] Late-onset SLE patients tend to have a more insidious onset of

disease and tend to have less major organ involvement and more benign disease course. [25] However, they have a poorer prognosis than patients who developed SLE before the age of 50 years, because of the generally higher frequency of comorbid diseases and higher organ damage, due to aging and longer exposure to "classical" vascular risk factors. [17,26,27].

## Aims of the Study:

To compare clinical and serological differences among juvenile, adult, and late-onset systemic lupus erythematosus in a cohort of SLE patients in our hospital.

## **Patients and Methods:**

#### Study design:

This study is a cross-sectional study

#### **Setting:**

This study will be conducted from January 2023 to January 2024 in Rheumatology Department, Sohag University Hospital. All the SLE patients visiting our department will be included in the study if they are fulfilling the inclusion criteria.

### **Inclusion criteria:**

- 1. Patients diagnosed as SLE according to SLICC 2012 or ACE/EULAR 2017 classification criteria.
- 2. Age (jSLE was defined as a diagnosis below the age of 18 years, and those diagnosed between 19 and 50 years of age were classified as aSLE (adult SLE), while ISLE (late onset SLE) was defined as a diagnosis at more than 50 years of age).
- 3. Patients with a disease duration of more than 6 months

#### **Exclusion criteria:**

1. Patients with had other autoimmune diseases, such as rheumatoid arthritis, systemic sclerosis, mixed connective tissue disease, overlap syndrom or primary Sjogren's syndrome, but not secondary Sjogren's syndrome or secondary antiphospholipid syndrome.

2. Patients who are not willing to be involved in the study

#### **Methods:**

All patients will be subjected to the following:

- 1. Thorough medical history of the patients
- 2. Full clinical examination including:
  - a. General examination and vital signs.
  - b. Complete rheumatological examination.
  - c. SLE disease activity index SLEDAI (ref).
  - d. SLICC damage index (ref).
- 3. Routine investigations (complete blood picture, erythrocyte sedimentation rate and liver functions).
- 4. Renal investigations:
  - a. Kidney functions
  - b. Urine analysis
  - c. 24 hours protein in urine and/or A/C ratio
  - d. Renal biopsy if indicated.
- 5. ANA test.
- 6. ANA profile for the most common 19 autoantibodies by immunoblot.

o Protocol

#### **Ethical considerations:**

- The study will be approved by the local Scientific Ethical Committee of the Faculty of Medicine, Sohag University.

- An informed written consent will be taken from all of the participants in the study after explaining the aim of the study.

#### **Statistical analysis:**

- Statistical package for social sciences (IBM-SPSS), version 24 (May 2016); IBM- Chicago, USA will be used for statistical data analysis.
- Data will be expressed as mean, standard deviation (SD), number and percentage. Mean and standard deviation will be used as descriptive value for quantitative data.
- Student t test will be used to compare the means between two groups, and one-way analysis of variance (ANOVA) test will be used to compare means of more than two groups. Mann Whitney test will be used instead of Student t test when the data are nonparametric.
- Pearson Chi square test will be used to compare percentages of qualitative variables, and Fisher exact test will be used instead of ordinary chi square test in cases of non-parametric data.
- Pearson correlation test will be used to compare two quantitative variables; and Spearman correlation test will be used instead if the data are non-parametric.
- For all these tests, the level of significance (P-value) can be explained as:
  - o No significance P > 0.05
  - o Significance P < 0.05
  - o High significance P < 0.001.

#### References

1 Von Feldt JM. Systemic lupus erythematosus. Recognizing its various

presentations. Postgrad Med 1995; 97: 79, 83, 86 passim.

- 2 Estes D, Christian CL. The natural history of systemic lupus erythematosus by prospective analysis. Medicine (Baltimore) 1971; 50: 85–95.
- 3 Fessler BJ, Boumpas DT. Severe major organ involvement in systemic

lupus erythematosus. Diagnosis and management. Rheum Dis Clin North Am 1995; 21: 81–98.

- 4 Borchers AT, Naguwa SM, Shoenfeld Y, Gershwin ME. The geoepidemiology of systemic lupus erythematosus. Autoimmun Rev 2010; 9: A277–A287.
- 5 Ferna' ndez M, Alarco' n GS, Calvo-Ale'n J, et al. A multiethnic, multicenter cohort of patients with systemic lupus erythematosus (SLE) as a model for the study of ethnic disparities in SLE. Arthritis Rheum 2007; 57: 576–584.
- 6 Arbuckle MR, James JA, Dennis GJ, et al. Rapid clinical progression
- to diagnosis among African-American men with systemic lupus erythematosus. Lupus 2003; 12: 99–106.
  - 7 Alarco' n GS, McGwin G Jr, Petri M, et al. Baseline characteristics of a multiethnic lupus cohort: PROFILE. Lupus 2002; 11: 95–101.
- 8 Alarco'n GS, McGwin G Jr, Roseman JM, et al. Systemic lupus erythematosus in three ethnic groups. XIX. Natural history of the accrual
- of the American College of Rheumatology criteria prior to the occurrence

of criteria diagnosis. Arthritis Rheum 2004; 51: 609-615.

9 Alarco' n GS, Calvo-Ale'n J, McGwin G Jr, et al. Systemic lupus erythematosus in a multiethnic cohort: LUMINA XXXV.

Predictive factors of high disease activity over time. Ann Rheum Dis 2006; 65: 1168–1174.

- 10 Alarco' n GS, McGwin G Jr, Bartolucci AA, et al. Systemic lupus erythematosus in three ethnic groups. IX. Differences in damage accrual. Arthritis Rheum 2001; 44: 2797–2806.
- 11 Uribe AG, Alarco' n GS. Ethnic disparities in patients with systemic

lupus erythematosus. Curr Rheumatol Rep 2003; 5: 364–369.

12 Samanta A, Feehally J, Roy S, Nichol FE, Sheldon PJ, Walls J. High prevalence of systemic disease and mortality in Asian subjects with systemic lupus erythematosus. Ann Rheum Dis 1991; 50:

Y Protocol

490-492.

13 Thumboo J, Uramoto K, O'Fallon WM, et al. A comparative study of the clinical manifestations of systemic lupus erythematosus in Caucasians in Rochester, Minnesota, and Chinese in Singapore, from 1980 to 1992. Arthritis Rheum 2001; 45: 494–500.

14 Richman IB, Taylor KE, Chung SA, et al. European genetic ancestry

is associated with a decreased risk of lupus nephritis. Arthritis Rheum 2012; 64: 3374–3382.

15 Isenberg D, Appel GB, Contreras G, et al. Influence of race/ethnicity

on response to lupus nephritis treatment: The ALMS study. Rheumatology 2010; 49: 128–140.

16 Tucker LB, Uribe AG, Ferna' ndez M, et al. Adolescent onset of lupus results in more aggressive disease and worse outcomes: Results of a nested matched case-control study within LUMINA, a multiethnic US cohort (LUMINA LVII). Lupus 2008; 17: 314–322.

- 17 Boddaert J, Huong DL, Amoura Z, Wechsler B, Godeau P, Piette JC. Late-onset systemic lupus erythematosus: A personal series of 47 patients and pooled analysis of 714 cases in the literature. Medicine (Baltimore) 2004; 83: 348–359.
- 18 Klein-Gitelman M, Reiff A, Silverman ED. Systemic lupus erythematosus in childhood. Rheum Dis Clin North Am 2002; 28: 561–577, vi–vii.
  - 19 Carren o L, Lo pez-Longo FJ, Monteagudo I, et al. Immunological and clinical differences between juvenile and adult onset of systemic lupus erythematosus. Lupus 1999; 8: 287–292.
- 20 Descloux E, Durieu I, Cochat P, et al. Influence of age at disease onset in the outcome of paediatric systemic lupus erythematosusRheumatology (Oxford) 2009; 48: 779–784.
- 21 Faco MM, Leone C, Campos LM, Febro<sup>^</sup> nio MV, Marques HH, Silva CA. Risk factors associated with the death of patients hospitalized

for juvenile systemic lupus erythematosus. Braz J Med Biol Res 2007; 40: 993–1002.

- 22 Hoffman IE, Lauwerys BR, De Keyser F, et al. Juvenile-onset systemic lupus erythematosus: Different clinical and serological pattern than adult-onset systemic lupus erythematosus. Ann Rheum Dis 2009; 68: 412–415.
- 23 Hersh AO, Trupin L, Yazdany J, et al. Childhood-onset disease as a predictor of mortality in an adult cohort of patients with systemic lupus erythematosus. Arthritis Care Res (Hoboken) 2010; 62:

A Protocol

1152-1159.

24 Moss KE, Ioannou Y, Sultan SM, Haq I, Isenberg DA. Outcome of a cohort of 300 patients with systemic lupus erythematosus attending a dedicated clinic for over two decades. Ann Rheum Dis 2002; 61: 409–413.

25 Formiga F, Moga I, Pac M, Mitjavila F, Rivera A, Pujol R. Mild presentation of systemic lupus erythematosus in elderly patients

## الملخص العربي

الذئبة الحمراء الجهازية (SLE) هو مرض مناعي ذاتي غير متجانس مع الاعراض ودورة متغيرة للغاية. يمكن أن يؤثر على كل عضو من أعضاء الجسم تقريبًا ويمكن ملاحظة العديد من الأعراض. يتم ملاحظة مثلا في الجلد والعضلات الهيكلية والدموية والمصلية بشكل شائع. [١] بعض المرضى يظهرون في الغالب اعراض دموية أو كلوية أو الجهاز العصبي المركزي. [٢٠٣]

قد يتميز المسار المرضى لمرض الذئبة الحمراء بفترات شفاء وانتكاسات مزمنة أو حادة. يمكن أن تؤثر عدة عوامل ، بما في ذلك العمر والعرق ، على طبيعة وشدة مرض الذئبة الحمراء ، كما تختلف الاستجابة للعلاج حسب العرق والعمر. يميل غير القوقازيين إلى الظهور بمرض حاد ، ومظاهر مرضيه أكثر حدة وتعددًا ، ونشاطًا أعلى للمرض. [٤-١٠] يُظهر ذوو الأصول الأسبانية والأفارقة والآسيويون اعتلال كلويًا ودمويًا ومصليًا وعصبيًا ومناعيًا أكثر تواترًا. علاوة على ذلك ، تختلف الاستجابة لعلاج التهاب الكلية الذئبي وفقًا للعرق. وبالمثل ، يمكن أن يؤثر العرق على طبيعة وشدة مرض الذئبة الحمراء واستجابته للعلاج: يؤثر سن البداية أيضًا على المظاهر المرضيه وشدة مرض الذئبة الحمراء. يعاني ما يقرب من ١٥-٠٠٪ من مرضى الذئبة الحمراء من ظهور المرض قبل سن البلوغ ، وحوالي ٢-٠٠٪ من جميع المرضى الذين يعانون من مرض الذئبة الحمراء يعانون من ظهور المرض بعد سن ٥٠. [١٦-١٨]

أفادت الدراسات أن مرضى الذئبة الحمراء في بداية الأحداث يميلون إلى أن يكون لديهم عرض ودورة أكثر عدوانية ، مع ارتفاع معدلات مشاركة الأعضاء وانخفاض متوسط العمر المتوقع من مرضى الذئبة الحمراء عند البالغين. [١٩-٢٤] يميل مرضى الذئبة الحمامية المجموعية المتأخرة إلى ظهور المرض بشكل أكثر حميدة. [٢٥] خداعًا ويميلون إلى مشاركة أعضاء رئيسية أقل ومسار مرضى أكثر حميدة. [٢٥]

) · Protocol

ومع ذلك ، فإن توقعات سير المرض لديهم أضعف من المرضى الذين أصيبوا بمرض الذئبة الحمراء قبل سن الخمسين ، بسبب التكرار الأعلى للأمراض المرضية المصاحبة وتلف الأعضاء بشكل أكبر ، بسبب الشيخوخة والتعرض لفترة أطول لمخاطر الأوعية الدموية "التقليدية" [٢٧،١٧،٢٦].

# أهداف الدراسة:

المقارنة بين الفروق الاكلينكايه والمعمليه بين مرض الذئبة الحمراء عند الأطفال ، والبالغين ، والذئبة الحمراءالمناعيه الجهازية المتأخرة في مجموعة من مرضى الذئبة الحمراء في مستشفانا.

# المرضى وطرق البحث:

# تصميم الدراسة:

هذه الدراسة عبارة عن دراسة مقطعية

# الضوابط:

ستجرى هذه الدراسة في الفترة من يناير ٢٠٢٣ إلى يناير ٢٠٢٤ في قسم أمراض الروماتيزم بمستشفى جامعة سوهاج سيتم ضم جميع مرضى الذئبه الحمراء الذين يزورون قسمنا في الدراسة إذا كانوا يستوفون معايير التضمين.

## معايير الاشتمال:

- 1. المرضى الذين تم تشخيصهم على أنهم مرضى الذئبه الحمراء وفقًا لمعاييرتصنيف ٢٠١٢.
- ۲. العمر (تم تعریف ذئبه حمراء فی الاطفال علی أنه تشخیص أقل من ۱۸
   عامًا ، بینما تم تصنیف الأشخاص الذین تم تشخیصهم بین ۱۹ و ۰۰ عامًا

على أنهم ذئبه حمراء في البالغين ، وتم تعريف ذئبه حمراء في كبار السن على أنه تشخيص عند أكثر من ٥٠ عامًا).

٣. المرضى الذين يعانون من المرض مدة تزيد عن ٦ أشهر.

## معايير الاستبعاد:

- المرضى الذين يعانون من أمراض المناعة الذاتية الأخرى ، مثل التهاب المفاصل الروماتويدي ، أو التصلب الجهازي ، أو متلازمة سجوجرن الأولية ، ولكن ليس متلازمة سجوجرن الثانوية أو متلازمة أضداد الشحوم الفوسفورية الثانوية.
  - ٢. المرضى الذين لا يرغبون في المشاركة في الدراسة

# وسوف يخضع جميع المرضى وحالات المراقبة لما يلي:

- ١. التاريخ الطبي الشامل من المرضى
  - ٢. الفحص الاكلينيكي بما في ذلك:
    - ١- الفحص العام
    - ٢- الفحص الروماتيزمي
- ٣. التحاليل الروتينية (صورة الدم كاملة، ومعدل الترسيب، وظائف الكبد وظائف الكلي).
  - ٤. قياس مضادات الأنوية.

# الإعتبار الأخلاقي:

- يتم الحصول على موافقة خطية من المريض بعد شرح هدف دراستنا.
- سيتم اعتماد بروتوكول الدراسة من قبل اللجنة الأخلاقية المحلية من كلية
   سوهاج للطب.



# جاه د قسم الرو

## جامعة سوهاج كلية الطب قسم الروماتيزم والتأهيل

المقارنة بين الفروق الاكلينيكيه والمعمليه بين مرض الذئبة الحمراء عند الأطفال ، والبالغين ، والذئبة الحمراءالمناعيه الجهازية المتأخرة

بروتوكول توطئة للحصول على درجة الدكتوراه في الطب الطبيعي والروماتيزم والتأهيل

# مقدمة من: ط. الاع محمد حمدان

مدرس مساعد بقسم الروماتيزم والتأهيل كلية الطب – جامعة سوهاج

تحت إشراف:

# د. عصام محمد أبو الفضل

أستاذ بقسم الروماتيزم والتأهيل كلية الطب – جامعة سوهاج

# د. حنان سید محمد ابو زید

استاذ مساعد بقسم الروماتيزم والتأهيل كلية الطب - جامعة سوهاج

> كلية الطب جامعة سوهاج ٢٠٢٢